CLINICAL TRIAL: NCT00022789
Title: Prevalence of Sleep Disordered Breathing in Children
Brief Title: Prevalence of Sleep-Disordered Breathing in Children
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Edward Bixler, Professor, Vice Chair Research, Milton S. Hershey Medical Center
Other Study IDs: 980; R01HL063772 (NIH)
Record Dates: First submitted 2001-08-14; First posted 2001-08-14 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Lung Diseases; Sleep Apnea Syndromes
Keywords: Sleep-Disordered Breathing
MeSH Terms: conditions — Lung Diseases; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

SUMMARY:
To investigate the prevalence and clinical significance of sleep-disordered breathing (SDB) in children.

DETAILED DESCRIPTION:
BACKGROUND:

SDB in children appears to be a common condition, affecting approximately 1 to 3 percent of children. Many aspects of childhood SDB remain understudied and poorly understood, including its precise prevalence, the optimal means of identifying children who should undergo polysomnography, and the potentially major impact of this condition on health, cognitive development, and behavior.

DESIGN NARRATIVE:

The population-based, cross-sectional study of 6- to 16-year-old schoolchildren in Dauphin County, Pennsylvania is a two-part study. In the first part of the study, parents of every child enrolled in local elementary schools will complete a questionnaire that will assess general sleep, behavior, and learning problems. In the second part of the study, 1,000 children will be randomly selected based on their risk for SDB, as determined by the questionnaire. They will be evaluated in a sleep laboratory to determine the presence of SDB. A thorough pediatric ear, nose, throat, and pulmonary evaluation will be conducted; school records and behavior will also be assessed. The parents of the children will be interviewed, and information will be collected on the family history of risk factors associated with childhood SDB. This strategy will be beneficial in establishing the prevalence and clinical significance of SDB in children.

ELIGIBILITY:
Inclusion Criteria:

* Phase I: Sampled all children by questionnaire completed by parent or guardian in three school districts in Dauphin County, Pennsylvania
* Phase II: Recruited a representative sample of 700 to complete a more detailed analysis in the laboratory

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Random representative population sample of children in elementary school (K-5)
Sampling Method: Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2001-08; Primary Completion 2006-06 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward O. Bixler, PhD, Study Chair — Milton S. Hershey Medical Center
Locations (1):
- Pennsylvania State University Hershey Medical Center, Hershey, Pennsylvania, United States